CLINICAL TRIAL: NCT04695873
Title: An Open-label, Randomised, Parallel-group, No-treatment Control Investigation to Determine the Effect of the Scholl Corn Foam Cushions, on Pain Levels When Used on Heloma Durum (Hard Corns) on the Dorsal Digital (Top of the Toe) and the Plantar Weight Bearing Areas (Ball of Foot) of the Feet
Brief Title: A 3 Day In-use Assessment of the Scholl Corn Foam Cushions on Pain Levels Associated With Heloma Durum.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Reckitt Benckiser Healthcare (UK) Limited (Industry)
Collaborators: O4 Research (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 4101101
Record Dates: First submitted 2021-01-04; First posted 2021-01-05 (Actual); Last update posted 2021-12-27 (Actual); Status verified 2021-12

CONDITIONS: Heloma Durum
Keywords: VAS Pain Assessment; Symptomatic Pain Relief
MeSH Terms: conditions — Callosities

STUDY DESIGN:
Intervention Model Description: An open label, randomized parallel group, no treatment control investigation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment Group (Experimental): Foam Cushion, applied daily on Days 1, 2 and 3 of the investigation.
  Interventions: Device: Corn Foam Cushion
- No Treatment Group (No Intervention): No treatment

INTERVENTIONS:
Device: Corn Foam Cushion — An anatomically shaped foam pad with a central hole. The upper layer is made from a honeycomb of interconnecting cells, the external facing surface is smooth, the underside is coated with adhesive.
  Arms: Treatment Group

SUMMARY:
This is an open-label, single-centre, parallel-group clinical investigation to evaluate the symptomatic pain relief, consumer acceptability and in-use tolerability of the Scholl Corn Foam Cushion in participants suffering from painful Heloma Durum over a 72-hour at home in-use period compared to a no-treatment control group.

DETAILED DESCRIPTION:
The investigation design will include an enrolment and randomisation visit followed by an at home in-use period and a final follow up phone call. The enrolment visit will include confirmation of eligibility and collection of baseline data, including baseline pain scores using the Visual Analogue Scale (VAS), medical history, demographics, and baseline Patient Reported Outcomes (PRO) assessments. Baseline data collected will be assessed to confirm eligibility before randomisation, first product application (treatment group only), initial pain (VAS) Participant Perceived Questionnaires (PPQ) and PRO assessments. During the at home in-use period, those participants randomised to the treatment group will reapply the product daily, complete pain assessments using the VAS (morning and evening), PPQs and PROs (Day 3 evening only). For participants randomised to the no-treatment group, they will complete pain assessments using the VAS (morning and evening) and PROs (Day 3 evening). All participants will continuously record Adverse Events (AE) and changes to concomitant medication throughout this period. During the follow up phone call, the participants will be contacted to establish any further AEs and/or changes to concomitant medication, additionally any queries related to diary entries will be made during this phone call. Participants will not need to return to the site unless advised to do so by the Principal Investigator (PI) or delegate.

After completion of the investigation, the Investigator will make an Assessment of Tolerance for each subject based on their pain scores (VAS), PPQ responses and AEs reported.

ELIGIBILITY:
Inclusion Criteria:

1. Participant has provided written informed consent.
2. Male or female participants aged: ≥ 18 and <70 years.
3. Otherwise healthy individual suffering from a single painful Heloma Durum on the dorsal digital or the plantar weight bearing area of the foot (or feet) as assessed by the Investigator or suitable delegate.
4. A baseline VAS score of ≥20 units and ≤75 units when measured on a VAS of 0-100.
5. Able to attend the investigation centre on the predefined day(s).
6. Owns or has access to a device with internet connectivity and is willing to download an investigation application and participate in the collection of patient-reported data (criterion only applicable for the use of electronic patient reported outcomes (ePRO) diary).
7. Is willing and capable of adhering to the investigational requirements.

Exclusion Criteria:

1. Individuals who have known allergies or sensitivities to latex, or any other ingredients of the product, which in the opinion of the Investigator is considered clinically relevant.
2. Individuals who have received any of the following treatment of their Heloma Durum:

   1. Conservative treatments (e.g. cushioning) within the last 2 days
   2. Chemical treatments (e.g. Salicylic Acid plaster) within the last 2 weeks
   3. Physical treatments (e.g. Heloma Durum debridement, including home debridement) within the last 6 weeks
3. Participants who, in the opinion of the Principal Investigator, have any unhealed skin at or surrounding the Heloma Durum as a result of any treatments used by the individual.
4. Significant foot deformities or inflammation (e.g. bunions, heel spurs, gout etc.).
5. Concurrent participation in another interventional clinical study/investigation, or participation within 30 days before Day 1 of this investigation.
6. Active infections of the foot or skin of the foot.
7. Those who are pregnant, attempting to become pregnant, or believe they may be pregnant or have given birth within the last 6 months (self-reported).
8. Participants who regularly use painkillers for ongoing conditions.
9. Participants who have taken over-the-counter painkillers within the last 2 days prior to screening.
10. Participants who are taking/or have taken prescription painkillers in the last 2 weeks prior to screening.
11. Participants who are unwilling to wear the same footwear throughout the investigation (footwear is defined as structured and enclosed shoes or trainers with a method of closure e.g. laces and a heel of less than 3 cm. Consistent wearing of socks/tights should be maintained throughout the investigation) for the duration of the investigation.
12. Any individuals with diabetes or poor blood circulation.
13. Any other callosity that is not identified as a Heloma Durum by a healthcare professional (i.e. soft corn, neurovascular corn, seed corn, fibrous corns).
14. Any Heloma Durum where the surrounding skin is inflamed or broken.
15. Any other features identified within the screening process that in the opinion of the Investigator will impact the safety or wellbeing of the participant or affect the outcome of the investigation.
16. Participants who are employees at the site or are a partner or first-degree relative of the Investigator.
17. Participants who fail to satisfy the Investigator of fitness to participate for any other reason

Ages: 18 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2021-06-16 (Actual); Primary Completion 2021-10-11 (Actual); Study Completion 2021-10-11 (Actual)

PRIMARY OUTCOMES:
Overall pain relief | Days 1-3
  Comparison of the average change from baseline in pain (VAS), across all timepoints from Day 1 to 3 between the treatment and no-treatment groups. The pain scores will be recorded on a pain visual analogue scale. which will be presented as a 0-100 scale with 0 indicating no pain at all and 100 indicating worst pain imaginable.

SECONDARY OUTCOMES:
Immediate pain relief | 25 minutes
  Comparison of change from baseline pain assessments (VAS) 25 minutes after replacing footwear between the treatment and no treatment groups. The pain VAS will be presented on a 0-100 scale with 0 indicating no pain at all and 100 indicating worst pain imaginable.
Specific Timepoint pain relief | Days 1-3
  Comparison of change from baseline in pain (VAS) at Day 1 evening, Day 2 morning and evening, Day 3 morning and evening following use of the Scholl Corn Foam Cushion whilst wearing footwear, between the treatment and no-treatment groups. The pain scores will be recorded on a pain visual analogue scale. which will be presented as a 0-100 scale with 0 indicating no pain at all and 100 indicating worst pain imaginable.
Percentage of participants experiencing a 25% pain reduction | Days 1-3
  Comparison of the percentage of participants who achieve 25% pain reduction from their baseline pain score at each time point between the treatment and no-treatment groups. The pain scores will be recorded on a pain visual analogue scale. which will be presented as a 0-100 scale with 0 indicating no pain at all and 100 indicating worst pain imaginable.
Consumer Acceptability | Days 1-3
  Participant Perceived Questionnaires at 25 minutes (+/- 5 minutes) after reapplication of footwear on day 1 and on the evening of Day 3, whilst wearing footwear (treatment group only).
Safety and Tolerability | Days 1-3
  Investigator Assessment of Tolerance for each participant in the treatment group only based on pain scores (VAS) and PPQ responses and AEs.
  Overall proportion of participants with Adverse Events / Adverse Device Effects (AEs/ADEs) i.e. the occurrence of one or more AEs/ADEs per participant.
Foot Health Improvement | Days 1-3
  Comparison of change in overall foot health from Baseline to Day 3, as assessed by the Podiatry Health Questionnaire (PHQ) Patient Reported Outcome (PRO) between the treatment and no-treatment groups.
Quality of Life Improvement | Days 1-3
  Comparison of change in overall quality of life from baseline to Day 3, as assessed by the EQ-5D-5L PRO between the treatment and no-treatment groups.

OTHER OUTCOMES:
Impact of Heloma Durum on work productivity and activity | Day 1
  Assessment of work productivity and activity impairment assessed by the Work Productivity and Activity Impairment: Specific Health Problem (WPAI:SHP) PRO.

CONTACTS AND LOCATIONS:
Overall Officials: David Watterson, Principal Investigator; Moneeb Saddiq, Study Director
Locations (1):
- Podiatry Services, West Community Services, Galway, Ireland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Becker BA, Childress MA. Common Foot Problems: Over-the-Counter Treatments and Home Care. Am Fam Physician. 2018 Sep 1;98(5):298-303. PMID 30216025
- [Background] Booth J, Mclnnes A. The aetiology and management of plantar callus formation. J Wound Care. 1997 Oct 2;6(9):427-430. doi: 10.12968/jowc.1997.6.9.427. PMID 27937673
- [Background] Burkhart CG. Skin disorders of the foot in active patients. Phys Sportsmed. 1999 Feb;27(2):88-101. doi: 10.3810/psm.1999.02.673. PMID 20086699
- [Background] Devlin NJ, Shah KK, Feng Y, Mulhern B, van Hout B. Valuing health-related quality of life: An EQ-5D-5L value set for England. Health Econ. 2018 Jan;27(1):7-22. doi: 10.1002/hec.3564. Epub 2017 Aug 22. PMID 28833869
- [Background] Dolan P. Modeling valuations for EuroQol health states. Med Care. 1997 Nov;35(11):1095-108. doi: 10.1097/00005650-199711000-00002. PMID 9366889
- [Background] Hodgkin SE, Hoffmann TJ, Ramsey ML. Minimizing Corns and Calluses. Phys Sportsmed. 1990 Jun;18(6):87-91. doi: 10.1080/00913847.1990.11710068. PMID 27452098
- [Background] Menz HB, Zammit GV, Munteanu SE. Plantar pressures are higher under callused regions of the foot in older people. Clin Exp Dermatol. 2007 Jul;32(4):375-80. doi: 10.1111/j.1365-2230.2007.02421.x. Epub 2007 Apr 8. PMID 17425648
- [Background] Omura EF, Rye B. Dermatologic disorders of the foot. Clin Sports Med. 1994 Oct;13(4):825-41. PMID 7805109
- [Background] Reilly MC, Zbrozek AS, Dukes EM. The validity and reproducibility of a work productivity and activity impairment instrument. Pharmacoeconomics. 1993 Nov;4(5):353-65. doi: 10.2165/00019053-199304050-00006. PMID 10146874
- [Background] Silfverskiold JP. Common foot problems. Relieving the pain of bunions, keratoses, corns, and calluses. Postgrad Med. 1991 Apr;89(5):183-8. doi: 10.1080/00325481.1991.11700901. PMID 1826149
- [Background] Rinaldi, F. & Clemente, F., 1994. The importance of formulation of a plaster containing salicylic acid in treatment of corns. Foot, The, 4(4), pp. 186-190.
- [Background] Grouios, 2004. Corns and calluses in athletes' feet: a cause for concern. Foot, The, 14(4), pp. 175-184.